CLINICAL TRIAL: NCT04716010
Title: Developing and Evaluating Product Messaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Wellcome Trust (Other); University of Edinburgh (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-3349; K01HL147713 (NIH)
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Results first posted 2022-09-09 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2021-08

CONDITIONS: Cancer of Colon; Cancer of Rectum
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Other): Products that contain red meat will not have warning labels or an increase in price.
  Interventions: Other: Control
- Warning Labels (Experimental): The warning labels are black octagons with white text that appear next to images of products that contain red meat. One label says "WARNING: Eating red meat contributes to colon and rectal cancer" and the other label says "WARNING: Eating red meat harms the environment."
  Interventions: Other: Warning Labels
- Tax (Experimental): The tax is a 30% increase in the price of products that contain red meat.
  Interventions: Other: Tax
- Combined Warning Labels and Tax (Experimental): The Combined Warning Labels and Tax arm features both the warning labels and tax. The warning labels are black octagons with white text that appear next to images of products that contain red meat. One label says "WARNING: Eating red meat contributes to colon and rectal cancer" and the other label says "WARNING: Eating red meat harms the environment." The tax is a 30% increase in the price of red meat products.
  Interventions: Other: Combined Warning Labels and Tax

INTERVENTIONS:
Other: Control — Participants will complete a shopping task in the online grocery store, and the products that contain red meat will not have warning labels or a 30% increase in price.
  Arms: Control
Other: Warning Labels — While completing the shopping task in the online grocery store, the health and environmental warning labels will appear next to the image of every product that contains red meat.
  Arms: Warning Labels
Other: Tax — While completing the shopping task in the online grocery store, all products containing red meat will have a 30% increase in price.
  Arms: Tax
Other: Combined Warning Labels and Tax — While completing the shopping task in the online grocery store, all products containing red meat will have the health and environmental warning labels appear next to the product image and a 30% increase in price.
  Arms: Combined Warning Labels and Tax

SUMMARY:
Purpose: To assess the impact of taxes, warnings, and a combination of taxes and warnings on US adults' decisions to purchase products that contain red meat in an online grocery store.

Procedures (methods): Participants will be recruited from Prime Panels (an online panel research company). Following online consent, participants will be assigned to one of four trial arms: 1) Control (no warning and no tax), 2) Warnings (all products that contain red meat have a health warning and environmental warning), 3) Tax (30% tax on products that contain red meat), and 4) Combined warning and tax (all products that contain red meat will have the two warnings and a 30% tax). Then, participant will enter an online grocery store reflecting their assigned arm. The participant will be instructed to complete a shopping task in the online grocery store. After completing the shopping task, participants will be redirected to an online survey and answer a series of questions about the shopping task, labels (excluding tax and control groups), and taxes (excluding warning and control groups). Questions will also include standard demographic and health related variables.

DETAILED DESCRIPTION:
Participants will be recruited from Prime Panels (an online panel research company). Following online consent, participants will be randomly assigned to one of four trial arms affecting the appearance of an online grocery store. Once in the online grocery store, participants will complete a shopping task. The participants will have 9 specified items to add to their shopping cart (1 pizza, 1 burrito, Burger patties [meat or vegetarian], Breakfast sausages [meat or vegetarian], 1 frozen individual meal, 1 loaf of bread, 1 sandwich filling [for example, ham, turkey, or peanut butter], 1 pack of tortillas, 1 taco filling [for example, steak, chicken, or beans]). Participants will be informed that they will not be spending any of their own money to complete the shopping task. After completing the shopping task, participants will be redirected to a survey. They will provide self-reported responses to survey questions (e.g. perceived healthfulness from eating red meat, perceived risk of cancer from eating red meat, thinking about the health/environmental harms of food products). Participants will also answer demographic and health related questions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Consumes red meat at least once per week.
* Responsible for at least 50% of grocery shopping for the household.
* Lives in the United States

Exclusion Criteria:

* Individuals who have participated in research studies from previous aims of this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4160 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey S Taillie, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Lindsay Jaacks, PhD, Principal Investigator — University of Edinburgh
Locations (1):
- Carolina Population Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A deidentified dataset and the survey codebook will be published to the Harvard Dataverse. The study protocol and statistical analysis plan will be published as supporting information with the study results in a peer-reviewed journal.
Supporting Information: Study Protocol, SAP
Time Frame: The deidentified dataset and corresponding survey codebook will be available upon publication of study results and will remain on the Harvard Dataverse indefinitely.
Access Criteria: Anyone who wishes to access the data.
URL: https://dataverse.harvard.edu/

REFERENCES:
- [Derived] Willits-Smith A, Taillie LS, Jaacks LM, Frank SM, Grummon AH. Effects of red meat taxes and warning labels on food groups selected in a randomized controlled trial. Int J Behav Nutr Phys Act. 2024 Apr 15;21(1):39. doi: 10.1186/s12966-024-01584-9. PMID 38622655
- [Derived] Taillie LS, Bercholz M, Prestemon CE, Higgins ICA, Grummon AH, Hall MG, Jaacks LM. Impact of taxes and warning labels on red meat purchases among US consumers: A randomized controlled trial. PLoS Med. 2023 Sep 18;20(9):e1004284. doi: 10.1371/journal.pmed.1004284. eCollection 2023 Sep. PMID 37721952

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Arm: Products that contain red meat will not have warning labels or an increase in price.
  Control: Participants will complete a shopping task in the online grocery store, and the products that contain red meat will not have warning labels or a 30% increase in price.
- Warning Labels Arm: The warning labels are black octagons with white text that appear next to images of products that contain red meat. One label says "WARNING: Eating red meat contributes to colon and rectal cancer" and the other label says "WARNING: Eating red meat harms the environment."
  Warning Labels: While completing the shopping task in the online grocery store, the health and environmental warning labels will appear next to the image of every product that contains red meat.
- Tax Arm: The tax is a 30% increase in the price of products that contain red meat.
  Tax: While completing the shopping task in the online grocery store, all products containing red meat will have a 30% increase in price.
- Combined Warning Labels and Tax Arm: The Combined Warning Labels and Tax arm features both the warning labels and tax. The warning labels are black octagons with white text that appear next to images of products that contain red meat. One label says "WARNING: Eating red meat contributes to colon and rectal cancer" and the other label says "WARNING: Eating red meat harms the environment." The tax is a 30% increase in the price of red meat products.
  Combined Warning Labels and Tax: While completing the shopping task in the online grocery store, all products containing red meat will have the health and environmental warning labels appear next to the product image and a 30% increase in price.
Period: Overall Study
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Started | 1039 | 1040 | 1039 | 1042
Completed | 887 | 891 | 874 | 866
Not Completed | 152 | 149 | 165 | 176

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm | Total
Number analyzed (Participants) | 887 | 891 | 874 | 866 | 3518
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (17.3) | 49.2 (17.7) | 50.1 (16.7) | 47.4 (17.2) | 48.8 (17.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Woman | 539 | 538 | 530 | 519 | 2126
  Man | 343 | 348 | 342 | 344 | 1377
  Non-binary | 3 | 5 | 2 | 3 | 13
  Self-described | 2 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Reporting of race/ethnicity was optional. Race and ethnicity were collected in separate survey questions. All reported data are included.
  Participants
    Hispanic (any race): number analyzed (Participants) | 879 | 886 | 866 | 859 | 3490
    Hispanic (any race) | 83 | 94 | 85 | 94 | 356
    Non-Hispanic White only: number analyzed (Participants) | 879 | 886 | 866 | 859 | 3490
    Non-Hispanic White only | 643 | 654 | 634 | 621 | 2552
    Non-Hispanic Black or African American only: number analyzed (Participants) | 879 | 886 | 866 | 859 | 3490
    Non-Hispanic Black or African American only | 80 | 87 | 76 | 89 | 332
    Non-Hispanic Asian or Pacific Islander only: number analyzed (Participants) | 879 | 886 | 866 | 859 | 3490
    Non-Hispanic Asian or Pacific Islander only | 33 | 29 | 38 | 31 | 131
    Non-Hispanic other race/multiracial: number analyzed (Participants) | 879 | 886 | 866 | 859 | 3490
    Non-Hispanic other race/multiracial | 40 | 22 | 33 | 24 | 119
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 887 | 891 | 874 | 866 | 3518

OUTCOME MEASURES:

1. Primary Outcome: Count of Products That Contain Red Meat
Description: The number of products in a participant's shopping basket that contain red meat.
Time Frame: At completion of ~15 minute shopping task
Measure: Mean (Standard Deviation); unit: red meat products
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 887 | 891 | 874 | 866
red meat products | 3.5 (1.7) | 3.2 (1.8) | 3.1 (1.6) | 2.7 (1.6)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p = 0.002, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p = 0.024, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is <0.05

2. Primary Outcome: Percentage of Red Meat Containing Products
Description: The percentage of products in a participant's shopping basket that contain red meat.
Time Frame: At completion of ~15 minute shopping task
Measure: Mean (Standard Deviation); unit: percentage of red meat items
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 887 | 891 | 874 | 866
percentage of red meat items | 39.0 (18.6) | 36.1 (19.8) | 34.0 (18.0) | 30.8 (18.5)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p = 0.001, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p = 0.022, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.001, Regression, Linear — The a priori threshold for statistical significance is <0.05

3. Secondary Outcome: Total Saturated Fat
Description: Total grams of saturated fat of products in a participant's shopping basket. This will be calculated by adding together the total saturated fat from each product in the participant's shopping basket. Saturated fat for each product will come from the product's nutrition facts panel. All products in the store are real life products that have designated nutrition facts panels.
Time Frame: At completion of ~15 minute shopping task
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 887 | 891 | 874 | 866
grams | 156.1 (91.9) | 156.1 (82.2) | 145.8 (78.6) | 143.4 (83.3)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is >0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

4. Secondary Outcome: Total Sodium
Description: Total grams of sodium of products in a participant's shopping basket. This will be calculated by adding together the total sodium from each product in the participant's shopping basket. Sodium for each product will come from the product's nutrition facts panel. All products in the store are real life products that have designated nutrition facts panels.
Time Frame: At completion of ~15 minute shopping task
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 887 | 891 | 874 | 866
grams | 18.5 (11.8) | 18.2 (7.0) | 17.9 (9.6) | 18.2 (12.0)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

5. Secondary Outcome: Total Calories
Description: Total calories of products in a participant's shopping basket. This will be calculated by adding together the total calories from each product in the participant's shopping basket. Calories for each product will come from the product's nutrition facts panel. All products in the store are real life products that have designated nutrition facts panels.
Time Frame: At completion of ~15 minute shopping task
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 887 | 891 | 874 | 866
kcal | 9844.4 (3098.0) | 10051.6 (3508.1) | 9661.1 (3151.8) | 9532.5 (2843.3)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

6. Secondary Outcome: Perceived Healthfulness
Description: Perceived healthfulness of eating red meat. Likert response options are on a 1 to 5 scale, with higher scores representing a higher perceived healthfulness of eating red meat.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for participants who provided response
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 884 | 887 | 868 | 866
Score on a scale | 3.3 (1.0) | 3.0 (1.1) | 3.3 (1.0) | 3.1 (1.0)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear

7. Secondary Outcome: Perceived Cancer Risk
Description: Perceived risk of colon and rectal cancer from eating red meat. Likert response options are on a 1 to 5 scale, with higher scores representing a higher perceived risk of colon and rectal cancer from eating red meat.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 884 | 887 | 869 | 866
Score on a scale | 2.8 (1.0) | 3.1 (1.1) | 2.7 (1.0) | 3.0 (1.1)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

8. Secondary Outcome: Perceived Environmental Risk
Description: Perceived risk of environmental harms from eating red meat. Likert response options are on a 1 to 5 scale, with higher scores representing a higher perceived risk of environmental harms from eating red meat.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 884 | 887 | 868 | 866
Score on a scale | 2.7 (1.1) | 2.8 (1.1) | 2.6 (1.0) | 2.8 (1.1)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

9. Secondary Outcome: Cognitive Elaboration (Health)
Description: Thinking about the health harms of food products while completing the shopping task. Likert response options are on a 1 to 5 scale, with higher scores representing a higher amount of thinking about health harms of food products.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 885 | 885 | 869 | 866
Score on a scale | 2.7 (1.3) | 2.8 (1.2) | 2.6 (1.2) | 2.8 (1.2)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

10. Secondary Outcome: Cognitive Elaboration (Environment)
Description: Thinking about the environmental harms of food products while completing the shopping task. Likert response options are on a 1 to 5 scale, with higher scores representing a higher amount of thinking about the environmental harms of food products.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 885 | 884 | 869 | 866
Score on a scale | 2.2 (1.2) | 2.4 (1.2) | 2.1 (1.1) | 2.4 (1.2)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

11. Secondary Outcome: Cognitive Elaboration (Price)
Description: Thinking about the price of food products while completing the shopping task. Likert response options are on a 1 to 5 scale, with higher scores representing a higher amount of thinking about the price of food products.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 885 | 887 | 869 | 866
Score on a scale | 4.1 (0.9) | 4.0 (0.9) | 4.1 (0.9) | 4.1 (0.9)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

12. Secondary Outcome: Specific Perceived Healthfulness
Description: Perceived healthfulness of specific red meat products (burgers, pepperoni pizza, and deli ham). Likert response options are on a 1 to 5 scale, with lower scores representing worse for health and higher scores representing better for health.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 884 | 887 | 868 | 866
Score on a scale | 2.9 (0.8) | 2.7 (0.9) | 2.9 (0.8) | 2.7 (0.9)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

13. Secondary Outcome: Specific Perceived Environmental Risk
Description: Perceived environmental harm of specific red meat products (burgers, pepperoni pizza, and deli ham). Likert response options are on a 1 to 5 scale, with lower scores representing worse for the environment and higher scores representing better for the environment.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 884 | 887 | 868 | 866
Score on a scale | 2.9 (0.7) | 2.7 (0.8) | 2.9 (0.7) | 2.8 (0.8)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

14. Secondary Outcome: Perceived Cost of the Burger Product.
Description: Perceived cost of the burger product. Likert response options are on a 1 to 5 scale, with lower scores representing less expensive and higher scores representing more expensive.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 878 | 886 | 868 | 860
score on a scale | 3.6 (0.9) | 3.6 (1.0) | 3.9 (0.9) | 3.9 (1.0)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

15. Secondary Outcome: Perceived Cost of the Pizza Product.
Description: Perceived cost of the pizza product. Likert response options are on a 1 to 5 scale, with lower scores representing less expensive and higher scores representing more expensive.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 881 | 887 | 868 | 860
score on a scale | 2.8 (1.0) | 2.8 (0.9) | 3.0 (0.9) | 3.0 (0.9)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

16. Secondary Outcome: Perceived Cost of the Ham Product.
Description: Perceived cost of the ham product. Likert response options are on a 1 to 5 scale, with lower scores representing less expensive and higher scores representing more expensive.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 881 | 886 | 868 | 859
score on a scale | 3.2 (0.9) | 3.2 (0.9) | 3.5 (1.0) | 3.5 (1.0)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

17. Secondary Outcome: Intention to Reduce
Description: Intention to reduce red meat consumption in the next 30 days. Likert response options are on a 1 to 5 scale, with higher scores representing a higher intention to reduce red meat consumption in the next 30 days.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 884 | 887 | 869 | 866
Score on a scale | 2.4 (1.2) | 2.5 (1.2) | 2.3 (1.1) | 2.5 (1.2)
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

18. Other Pre Specified Outcome: Percentage of Participants Who Support Tax
Description: Support of policy for taxes on red meat products in the U.S. Likert response options are on a 1 to 5 scale, with higher scores representing a greater deal of support. Those who indicated '4' or '5' were assumed to more strongly agree to support a red meat product tax. This measure reports the percentage of those with a response of '4' or '5'.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response
Measure: Number; unit: percentage of participants
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 883 | 887 | 869 | 863
percentage of participants | 21.40 | 22.44 | 15.77 | 21.78
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

19. Other Pre Specified Outcome: Percentage of Participants Who Support Health Warning Label
Description: Support of policy for health warning labels on red meat products in the U.S. Likert response options are on a 1 to 5 scale, with higher scores representing a greater deal of support. Those who indicated '4' or '5' were assumed to more strongly agree to support a health warning label. This measure reports the percentage of those with a response of '4' or '5'.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response
Measure: Number; unit: percentage of participants
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 883 | 887 | 869 | 863
percentage of participants | 42.13 | 49.38 | 37.86 | 48.44
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

20. Other Pre Specified Outcome: Percentage of Participants Who Support Environmental Warning Label
Description: Support of policy for environmental warning labels on red meat products in the U.S. Likert response options are on a 1 to 5 scale, with higher scores representing a greater deal of support. Support of policy for taxes on environmental warning labels in the U.S. Likert response options are on a 1 to 5 scale, with higher scores representing a greater deal of support. Those who indicated '4' or '5' were assumed to more strongly agree to support an environmental warning label. This measure reports the percentage of participants with a response of '4' or '5'.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response
Measure: Number; unit: percentage of participants
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 883 | 887 | 869 | 863
percentage of participants | 40.20 | 44.87 | 33.14 | 44.26
Statistical Analysis 1: Comparison: Control Arm vs Warning Labels Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 2: Comparison: Control Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 3: Comparison: Control Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 4: Comparison: Warning Labels Arm vs Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 5: Comparison: Warning Labels Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p > 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05
Statistical Analysis 6: Comparison: Tax Arm vs Combined Warning Labels and Tax Arm; Test type: Superiority; p < 0.05, Regression, Linear — The a priori threshold for statistical significance is <0.05

21. Other Pre Specified Outcome: Mean Modified Waterlander Acceptability Scale Score
Description: Acceptability of the online grocery store. Likert response options are on a 1 to 5 scale, with higher scores representing a higher amount of agreement.
  Acceptability of the online grocery store is measured using 3 items adapted from Waterlander et al., 2011. Responses to the 3 items will be averaged to create an acceptability score sum ranging from 3-15 then divided by the total number of questions asked (n = 3).
  Prompt: Say whether you agree or disagree with the following statements.
  I could easily find all of the food and beverages I was looking for in the online grocery store.
  There were enough food and beverage options in the online grocery store.
  This online grocery store felt like a real online grocery store.
  Waterlander WE, Scarpa M, Lentz D, Steenhuis IHM. The virtual supermarket: an innovative research tool to study consumer food purchasing behavior. 2011;11:589. DOI: 10.1186/1471-2458-11-589.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 885 | 889 | 869 | 866
Score on a scale | 4.1 (0.8) | 4.0 (0.9) | 4.1 (0.8) | 4.0 (0.9)

22. Other Pre Specified Outcome: Ease of Store Use
Description: Ease of use of the online grocery store. Likert response options are on a 1 to 5 scale, with higher scores representing more agreement that the online grocery store is easy to use.
Time Frame: ~15 minutes post-test computer survey following the ~15 minute shopping task
Population: Assessed for all participants who provided response
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
Number analyzed (Participants) | 885 | 889 | 869 | 865
Score on a scale | 4.1 (0.9) | 4.0 (1.0) | 4.1 (0.9) | 4.1 (0.9)

ADVERSE EVENTS:
Time Frame: From the time of signing the Informed Consent and completion of the shopping task (~15 minutes) through completion of the post-shopping task computer survey (~15 minutes), an approximate total of up to 30 minutes.
Arm/Group | Control Arm | Warning Labels Arm | Tax Arm | Combined Warning Labels and Tax Arm
All-Cause Mortality (participants affected / at risk) | 0/887 | 0/891 | 0/874 | 0/866
Serious Adverse Events (participants affected / at risk) | 0/887 | 0/891 | 0/874 | 0/866
Other Adverse Events (participants affected / at risk) | 0/887 | 0/891 | 0/874 | 0/866

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT04716010/Prot_004.pdf
  • Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT04716010/SAP_003.pdf